CLINICAL TRIAL: NCT02279602
Title: Rollover for Study OX4218s, A P2 Study to Investigate Safety and Activity of Fosbretabulin Tromethamine in the Treatment of Well-Differentiated, Low-to-Intermediate-Grade Unresectable, Recurrent or Metastatic PNET or GI-NET With Elevated Biomarkers
Brief Title: Rollover Protocol for Subjects Who Have Responded on Study 4218s - A Phase 2 Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mateon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OX4219s
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Neuroendocrine Tumors
Keywords: Pancreatic; Gastrointestional
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — fosbretabulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Subjects will receive fosbretabulin at the same dose and frequency as in study OX4218s
  Interventions: Drug: fosbretabulin

INTERVENTIONS:
Drug: fosbretabulin — fosbretabullin, 60 mg/m2 weekly for up to 1 year
  Other Names: CA4P, combretastatin A-4 phosphate

SUMMARY:
Subjects achieving a clinical response in study OX4218s with a biomarker reduction or symptom response are eligible to enroll in this rollover study to continue once every three weeks fosbretabulin infusions for up to one year.

DETAILED DESCRIPTION:
Subjects enrolled in the PNET/GI-NET study OX4218s received weekly dosing with fosbretabulin for up to 3 cycles or approximately 9 weeks. Subjects achieving a clinical response with a biomarker reduction or symptom response based on investigator assessment are eligible to enroll in this rollover study (protocol OX4219s). Subjects will receive fosbretabulin every three weeks for a maximum of approximately one year or until disease progression, unacceptable toxicity, consent withdrawal, protocol-noncompliance, or the investigator feels that it is no longer in the subject's best interest to continue therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been treated in the OXiGENE-sponsored Phase 2 study OX4218s

Exclusion Criteria:

* Subject has not received fosbretabulin treatment in the study OX4218s

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in biomarkers from baseline | 48 Weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford University School of Medicine, Stanford, California
  - Markey Cancer Center, Clinical Research Office, Lexington, Kentucky
  - Montefiore, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Froedtert Hospital, Medicial College of Wisconsin, Milwaukee, Wisconsin